CLINICAL TRIAL: NCT00000849
Title: Phase I/II Trial of Recombinant Interleukin-2 In Symptomatic Human Immunodeficiency Virus-Infected Children
Brief Title: A Study to Test the Safety of Recombinant Interleukin-2 (rIL-2) in HIV-Infected Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: ACTG 299; 11275 (Registry Identifier: DAIDS ES Registry Number); PACTG 299
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-29 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Interleukin-2; Immunity, Cellular; Dose-Response Relationship, Drug; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Viral Load
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — aldesleukin

INTERVENTIONS:
Drug: Aldesleukin

SUMMARY:
The purpose of this study is to determine the safety and maximum tolerated dose (the highest dose that can be given safely) of recombinant Interleukin-2 (rIL-2) in HIV-infected children. This study also evaluates the effect of rIL-2 on the immune system of these patients.

IL-2 is a substance naturally produced by the body's white blood cells that plays an important role in helping the body fight infection. HIV-infected patients do not produce enough IL-2, and it is hoped that the use of rIL-2 may improve immune system function in these patients. First, it is necessary to determine the safety and effectiveness of this drug in HIV-infected children.

DETAILED DESCRIPTION:
According to study records, IL-2 has not been tested in HIV-infected children. Experience with IL-2 in pediatric populations is extremely limited. Pahwa et al. gave 30,000 units/kg daily IV to a child with severe combined immunodeficiency. This dose was well tolerated and the patient improved clinically as well as immunologically. Part A is necessary to determine the maximum tolerated dose of IL-2 in infected children. Part B will determine the efficacy of the maximum tolerated dose in infected children.

Part A: Children will receive rIL-2 intravenously for 5 days every 8 weeks for 3 cycles. The study will enroll 4 patients in each of 3 dose levels. Dose escalation may occur if all 4 patients in a dose level tolerate therapy without evidence of Grade 3 (or higher) toxicity. If 1 of 4 subjects in any dose level experiences at least Grade 3 toxicity, 2 additional patients will be enrolled in that dose level. If 1 of these 2 additional patients experiences at least Grade 3 toxicity, dose escalation will not proceed. NOTE: Once Part A is completed and the maximum tolerated dose is established, children who participated in Part A and received less than the maximum tolerated dose will be offered additional therapy consisting of 3 cycles of rIL-2 at the maximum tolerated dose.

Part B: Children will receive rIL-2 intravenously at the maximum tolerated dose established in part A. Treatment will be given for 5 days every 8 weeks for 3 cycles. [AS PER AMENDMENT 6/4/98: Children will receive rIL-2 intravenously at the lowest dose for 5 days every 8 weeks for 6 cycles. Patients who received this dose in part A will also be offered this regimen.]

ELIGIBILITY:
Inclusion Criteria

Children may be eligible for this study if they:

* Are HIV-positive.
* Have decreased immune system functioning (CD4 count 500-1000 for 3- to 5-year-olds or CD4 count 200-500 for 6- to 12-year-olds).
* Have symptomatic HIV infection.
* Have a viral level less than 400 copies/ml.
* Are between the ages of 3 and 12 (consent of parent or guardian required).

Exclusion Criteria

Children will not be eligible for this study if they:

* Have an active opportunistic infection.
* Are pregnant.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27
Dates: Study Completion 2001-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Starr, Study Chair; Steven Douglas, Study Chair
Locations (14):
- United States (14):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - UCSF Pediatric AIDS CRS, San Francisco, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - Texas Children's Hosp. CRS, Houston, Texas
  - VCU Health Systems, Dept. of Peds, Richmond, Virginia

REFERENCES:
- [Background] Zeng C, Mawhinney S, Baron AE, McFarland EJ. Evaluating ELISPOT summary measures with criteria for obtaining reliable estimates. J Immunol Methods. 2005 Feb;297(1-2):97-108. doi: 10.1016/j.jim.2004.12.006. PMID 15777934